CLINICAL TRIAL: NCT04629755
Title: A Smartphone Intervention for Relational and Mental Well Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jonathan Kanter, Research Associate Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009897
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Depression; Loneliness; Relation, Interpersonal; Covid19
MeSH Terms: conditions — Depression; COVID-19 | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention was delivered via a series of daily text messages to mobile phones. Participants first were delivered an introductory text message at 6:00 pm on Day 7 of the study. This message alerted the participants to expect their first suggestion via text message at 8:00 am the following morning. For the next 14 days (Days 8 - 22), participants received one of 14 suggestions in random order. The specific daily suggestions varied in length and complexity: The simplest ones included text messages and a brief audiofile delivered via text; the more complex suggestions included text messages and a link to a web-page, which included text or embedded audiofiles describing why a suggestion was being made, how to engage in the suggested practice, and audiotaped exchanges between members of the production team describing what it was like to try the practices themselves. Some suggestions were supplemented with additional reminder and check-in text messages at noon and 4:00 pm.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Assessment only.

INTERVENTIONS:
Behavioral: Intervention — The intervention was delivered via daily text messages to mobile phones during two weeks in the midst of the Covid-19 pandemic. Each message provided a link to a brief suggestion for an action or actions to take each day to improve relational closeness and well-being. Critical to the rationale for this intervention was the position that relationship science has developed key insights into what works and does not work to build and maintain closeness. These insights could be translated into brief and effective suggestions that individuals could implement daily, thereby quickly improving relational well-being and decreasing depression and loneliness at a critical time.
  Arms: Intervention

SUMMARY:
The primary aim of this study is to provide and evaluate a phone-based intervention to improve relational and mental well-being during the COVID-19 crisis. This information also will help us understand how individuals are responding to COVID-19 and have the potential to inform psychological and policy level interventions.

DETAILED DESCRIPTION:
We conducted a randomized intervention trial of a mobile-based intervention that offered participants daily suggestions for 14 days on how to improve relational and mental well-being during the COVID-19 pandemic. A sample of 1765 adults residing in the United States participated in the study and were assigned to control or intervention conditions. To measure outcomes, all participants received a daily text message to their smartphones every evening for 28 days linking to a survey on relational and mental well-being. Participants also received a survey link on Days 56 and 72. Intervention participants received additional text messages in the mornings of Days 7 - 22 presenting the intervention suggestions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Resides in United States
* Possesses smartphone
* Willing to share phone number and email to researchers

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1765 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Change in depressed mood | Measured every evening for 28 days; the first 6 days constituted baseline measurement; change was assessed over Days 7 - 28 with baseline as a covariate
  Depressed mood was measured using the first two symptom items of the Patient Health Questionnaire-2, "I felt down, depressed, or hopeless today" and "I had little interest or pleasure in doing things today"; both were rated with a slider from 0 (None of the time) to 10 (All of the time) with anchors "Some of the time" and "Most of the time" spaced evenly between.
Change in loneliness | Measured every evening for 28 days; the first 6 days constituted baseline measurement; change was assessed over Days 7 - 28 with baseline as a covariate
  Loneliness was measured using two items adapted from the UCLA Loneliness Scale, "I felt lonely today" and "I felt left out today" using a slider from 0 (Not at all) to 10 (Extremely).
Change in relationship quality | Measured every evening for 28 days; the first 6 days constituted baseline measurement; change was assessed over Days 7 - 28 with baseline as a covariate
  Relationship quality was measured using two items, "I felt closer and more connected to important people in my life today" with a slider including 0 (Not at all), 5 (A moderate amount) and 10 (Very much so) and "I felt satisfied with my relationships today" with a slider from 0 (Not at all) to 10 (Extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Kanter, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided